CLINICAL TRIAL: NCT01421719
Title: Onabotulinum Toxin Type A (BTX-A) For Treatment of Neurogenic Overactive Bladder Due to Parkinson's Disease: Safety and Efficacy
Brief Title: Safety and Efficacy of botulinumA Toxin (BotoxA) for Treatment of Neurogenic Bladder of Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Rodney U Anderson, Professor of Urology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000124
Record Dates: First submitted 2011-08-19; First posted 2011-08-23 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Parkinson's Disease; Neurogenic Bladder; Urinary Incontinence; Clostridium Botulinum Toxin Adverse Reaction
Keywords: Parkinson's Disease; Neurogenic Bladder; Urinary Incontinence; botulinum toxin; cystoscopy; Effect of Other Parasympatholytics [Anticholinergics and Antimuscarinics] and Spasmolytics
MeSH Terms: conditions — Parkinson Disease; Urinary Bladder, Neurogenic; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- botulinum toxin treatment (Experimental): botulinum toxin treatment Injection of Botox into urinary bladder for neurogenic symptoms.
  Interventions: Drug: Cystoscopic injection of Botox into the urinary bladder

INTERVENTIONS:
Drug: Cystoscopic injection of Botox into the urinary bladder — 100 U of Botox A injected transurethrally into the urinary bladder muscle and submucosa.
  Other Names: Botox A (Allergan, Inc)

SUMMARY:
The basic nerve deficit of Parkinson's disease (PD) leads to lower urinary tract symptoms of frequency, urgency and urge urinary incontinence. Lower urinary tract symptoms tend to occur at more advanced stages of PD. In the over-65 year old age group, where 1% of men suffer from this disease, they are also prone to development of benign prostatic hyperplasia (BPH) and consequent associated lower urinary tract dysfunction. Similarly the over 65-year age group develop spontaneous overactive bladder up to a prevalence of 30% of both men and women. The urologic disorder is exceedingly devastating in reducing the quality of life in these individuals due to the lower urinary tract symptoms and ultimate urinary incontinence in a high proportion of patients.

While attempts at pharmacologic treatment are partially satisfactory many patients are intolerant of oral drugs.

Botulinum-A neurotoxin (BTX-A) has been shown in pilot trials to be quite effective in reducing overactive bladder symptoms and is specifically beneficial for a wide-variety of neurogenic bladder causes of over activity . The treatment procedure of injecting the detrusor muscle of the bladder with BTX-A is quite simple, does not impose significant risks to the patient, and can be performed as an office urologic procedure.

This pilot clinical trial intends to demonstrate the safety and efficacy of low-dose Botox-A injections into the bladder to improve urinary symptoms in 20 patients.

DETAILED DESCRIPTION:
This open-label pilot study will evaluate the safety and efficacy of intra-detrusor injections of botulinum-A toxin (BTX-A) in 20 male or female patients with Parkinson's disease and neurogenic overactive bladder with or without urinary incontinence, but without evidence of significant urinary retention (>25% of bladder capacity at void).

Patients will be invited to participate based upon subjective symptoms of uncontrolled lower urinary tract urgency, frequency and urinary incontinence. Only patients who have a Hoehn and Yahr Stage IV or better (or UPDRS equivalent) will be considered. Patients must have tried anti-muscarinic agents and failed to improve or were intolerant of these pharmacologic agents. Oral anti-muscarinic medications will be discontinued two weeks prior to urodynamics testing and treatment visit. At baseline urinary symptom scores will be obtained using The King's Health Questionnaire (KHQ, a validated scoring system for urinary symptoms) and the AUA Urinary Symptom Score. In addition a 3-day fluid intake and urinary outflow timed voiding diary will be submitted at the time of testing and treatment as well as follow-up visits.

After signing an informed consent and meeting all inclusion and exclusion criteria, patients will be tested with urodynamic studies to determine current lower urinary tract neurophysiologic functioning. A "free-flow" urinary flow rate and post-void residual urine volume test will be performed as well as filling cystometrogram and pressure/flow measurement. Patients with evidence of outlet obstruction (high pressure/low flow) will be excluded from the study. Only patients with a post-void residual urine volume less than or equal to 25% of the total bladder volume at void will be included. No catheters or other measurement devices will be attached to the body at the time of the initial free urinary flow and post-void urine volume measurement. A repeat pressure/flow determination will be performed during the urodynamics cystometrogram.

After qualification to proceed, patients will then be transferred to the adjoining cystoscopy suite. Pre-procedure oral sedation and analgesia will be given. Subjects will undergo cystoscopy under topical lidocaine anesthesia and undergo 25-gauge needle injections of BTX-A. BTX-A treatment for each participant will be limited to a total dose of 100 units in a minimum of 10 to 20 locations. Any patient unable to void after the procedure will receive an indwelling catheter for 24 hours. Patients will be contacted by telephone within 24-48 hours after the procedure for safety assessment. Follow-up clinic visit evaluations will occur at 1 month, 3 months, 6 months and 9 months. A 3-day voiding diary, King's Health Questionnaire, AUA Symptom Score sheet and Global Response Assessment (GRA) Questionnaire will be collected at each follow-up visit. Incontinence will be documented on this diary. Uroflowmetry and post-void residual volume will also be assessed at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:•

* Male or female subjects, 50 to 85 years of age.
* Patients diagnosed with Parkinson's disease prior to lower urinary tract symptoms.
* Documentation of low volume desire to void and/or unstable detrusor contractions with or without incontinence on cystometrogram. Voiding diary consistent with overactive bladder
* Written informed consent has been obtained.
* Ability to follow study instructions and likely to complete all required visits.
* Written authorization for Use and Release of Health and Research Study Information has been obtained.
* Subject has minimum to moderate severity/stage of disease, Hoehn and Yahr stage IV or less (or UPDRS equivalent)
* Usual and customary medications allowed

Exclusion Criteria:

* Uncontrolled clinically significant medical condition other than the condition under evaluation
* Known allergy or sensitivity to any of the components in the study medication.
* Concurrent participation in another investigational drug or device study or participation within 60 days period of time prior to study
* New anticholinergic medication. Should discontinue any anti-muscarinic medication 14 days prior to injection.
* Treatment with botulinum toxin of any serotype prior to enrollment in study (if applicable).
* Any medical condition that may put the subject at increased risk with exposure to BTX-A including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other disorder that might interfere with neuromuscular function (if applicable).
* Evidence of alcohol, drug abuse or other relevant neuropsychiatric condition (if applicable)
* Urinary tract infection
* Significant BPH with evidence of severe bladder trabeculation
* Greater than 50% post-void residual urine volume
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodney U Anderson, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Hospital and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period extended between February 1, 2009 and September 2010. Stanford University Clinics represented location for enrollment and clinical trial.
Pre-assignment Details: Patients underwent screening in the clinic and were excluded per protocol prior to enrollment. Open label study.
Groups:
- Botulinum Toxin Treatment: Injection of Botox into urinary bladder for neurogenic symptoms.
Period: Overall Study
Arm/Group | Botulinum Toxin Treatment
Started | 20
Completed | 16
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Botulinum Toxin Treatment
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.95 (8.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Secondary Outcome: Number of Incontinence Episodes Per Day
Description: Urinary incontinence 6 months after treatment (n=16). Data are included for participants who completed all diary entries and attended the Month 6 visit
Time Frame: 6 months
Population: Per protocol. Quantified from 3-day voiding diary at baseline and each clinical evaluation to 6 months. Mean change in daily incontinence made up analysis.
Measure: Mean (Standard Deviation); unit: leaks/day
Groups:
- Urinary Leaks Per Day: 3-day voiding diary produced the clinical observation as an average per evaluation milestone.
Arm/Group | Urinary Leaks Per Day
Number analyzed (Participants) | 16
leaks/day
  Baseline urinary incontinence | 3.76 (2.57)
  Urinary incontinence 6 months after treatment | 1.40 (1.43)
Statistical Analysis 1: Comparison: Urinary Leaks Per Day; Paired t test comparison of baseline number of urinary leaks per day versus number of leaks per day at 6 month evaluation after treatment; Test type: Superiority or Other; p = 0.0087, t-test, 2 sided

2. Primary Outcome: Number of Patients Requiring Catheterization for Urinary Retention Secondary to Treatment.
Description: Requirement for catheter because of urinary retention.
Time Frame: zero to six months
Measure: Number; unit: participants
Arm/Group | Botulinum Toxin Treatment
Number analyzed (Participants) | 20
participants | 0

ADVERSE EVENTS:
Time Frame: 0 to 6 months.
Description: Primary consideration of adverse events included pain, bleeding, infection and urinary retention.
Arm/Group | Botulinum Toxin Treatment
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botulinum Toxin Treatment (N=20)
urinary tract infection (Renal and urinary disorders) | 1 (1) — Any urinary tract infection occurring within 30 days of injection procedure

LIMITATIONS AND CAVEATS:
The limitations of this trial involved the primary disease disorder of Parkinson's Disease and difficulty of communication with subjects; Four patients withdrew from the study prior to the 6-month endpoint because of loss of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No